CLINICAL TRIAL: NCT04308174
Title: Randomized Phase 2 Study of Preoperative Gemcitabine Plus Cisplatin With or Without Durvalumab (MEDI4736) Followed by Postoperative Durvalumab (MEDI4736) in Patients With Localized Biliary Tract Cancer
Brief Title: Neoadjuvant Gemcitabine Plus Cisplatin With or Without Durvalumab in Resectable Biliary Tract Cancer
Acronym: DEBATE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Changhoon Yoo, Assistant professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESR-18-14059
Record Dates: First submitted 2020-03-12; First posted 2020-03-13 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Biliary Tract Neoplasms; Gallbladder Cancer; Cholangiocarcinoma
Keywords: Biliary tract cancer; Immunotherapy; Neoadjuvant chemotherapy
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms; Cholangiocarcinoma | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Durvalumab + Gem/Cis (Experimental): <Investigational arm: preoperative phase (up to 4 cycles)> Durvalumab 1,500 mg IV on Day 1, every 3 weeks (preop period) 1,500 mg IV Day 1, every 4 weeks (postop period) Gemcitabine 1,000 mg IV on Day 1 and 8, every 3 weeks Cisplatin 25 mg IV on Day 1 and 8, every 3 weeks
  <Postoperative therapy for all patients (up to 6 cycles)> Durvalumab 1,500 mg IV Day 1, every 4 weeks (postop period)
  Interventions: Drug: Durvalumab + Gem/Cis
- Gem/Cis (Active Comparator): <Control arm: preoperative phase (up to 4 cycles)> Gemcitabine 1,000 mg IV on Day 1 and 8, every 3 weeks Cisplatin 25 mg IV on Day 1 and 8, every 3 weeks
  <Postoperative therapy for all patients (up to 6 cycles)> Durvalumab 1,500 mg IV Day 1, every 4 weeks (postop period)
  Interventions: Drug: Gem/Cis

INTERVENTIONS:
Drug: Durvalumab + Gem/Cis — Neoadjuvant Durvalumab + Gemcitabine/Cisplatin
  Arms: Durvalumab + Gem/Cis
Drug: Gem/Cis — Neoadjuvant Gemcitabine/Cisplatin
  Arms: Gem/Cis

SUMMARY:
Considering that the poor prognosis of resected biliary tract cancer and negative impact on the survival outcomes of R1/R2 resection, neoadjuvant chemotherapy may improve R0 resection rates and the survival outcomes of patients with resectable biliary tract cancer. The addition of durvalumab to gemcitabine/cisplatin as neoadjuvant chemotherapy may improve the R0 resection rates compared to gemcitabine/cisplatin in patients with localized biliary tract cancer. In this phase 2 trial, a total of 45 patients with localized biliary tract cancer will be 2:1 randomized to durvalumab plus gemcitabine/cisplatin or gemcitabine/cisplatin.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
* Age > 19 years at time of study entry
* Histologically confirmed adenocarcinoma of biliary tract (intrahepatic, hilar or extrahepatic cholangiocarcinoma, or gallbladder carcinoma).
* Localized, potentially resectable, non-metastatic disease (determined at the discretion of attending surgeons) based on the results of CT, MRI or PET-CT scans.
* No active uncontrolled infection, except chronic viral hepatitis under antiviral therapy.
* Eastern Cooperative Oncology Group (ECOG performance status of 0 or 1
* Body weight >30kg
* Adequate normal organ and marrow function
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* No other malignant disease apart from non-melanotic skin cancer, carcinoma in situ of the uterine cervix, localized prostate or papillary thyroid cancer, or any other cancer where treated with curative intent > 5 years previously without evidence of relapse

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent or to complete the protocol or a history of non-compliance
* Obstruction of gastrointestinal tract
* Active gastrointestinal bleeding
* Myocardial infarction within 6 months prior to the study medication, and other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension)
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardise compliance with the protocol
* Combined hepatocellular carcinoma/cholangiocarcinoma is excluded.
* History of allogenic organ transplantation.
* History of another primary malignancy except for

  1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  3. Adequately treated carcinoma in situ without evidence of disease
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart).
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
* Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Ro resection rate | 4 months
  Surgical resection without any residual cancer

SECONDARY OUTCOMES:
Overall survival | 1 year
  Time between the start of study treatment and any cause of death
Event-free survival | 1 year
  Time between the start of study treatment and disease progression or any cause of death
Adverse events | 13 months
  Number of patients experiencing adverse events graded by National Cancer Institute Common Terminology Criteria version 5
Response rate | 4 months
  Graded by Response Evaluation Criteria in Solid Tumors version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Changhoon Yoo, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be determined at the time of completion of the study.

REFERENCES:
- [Background] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Background] Kang J, Jeong JH, Hwang HS, Lee SS, Park DH, Oh DW, Song TJ, Kim KH, Hwang S, Hwang DW, Kim SC, Park JH, Hong SM, Kim KP, Ryoo BY, Yoo C. Efficacy and Safety of Pembrolizumab in Patients with Refractory Advanced Biliary Tract Cancer: Tumor Proportion Score as a Potential Biomarker for Response. Cancer Res Treat. 2020 Apr;52(2):594-603. doi: 10.4143/crt.2019.493. Epub 2019 Dec 18. PMID 32019287
- [Background] Valle JW, Borbath I, Khan SA, Huguet F, Gruenberger T, Arnold D; ESMO Guidelines Committee. Biliary cancer: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2016 Sep;27(suppl 5):v28-v37. doi: 10.1093/annonc/mdw324. No abstract available. PMID 27664259